CLINICAL TRIAL: NCT02738424
Title: Reproductibility of Lumbar Spine ADC Based on Different Post-processing Softwares
Acronym: ADC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN642015/CHUSTE
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; MRI
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 3T patients : Calculate the ADC scores: In this group all the patients perform a 3 Tesla RMI. With these data, three methods will be used to calculate the ADC score : Siemens, PACS (picture archiving and communication system) Carestream, Osirix. The ADC scores obtained with these three post-processing softwares will be compared.
  Interventions: Other: Calculate the ADC scores
- 1.5T patients : Calculate the ADC scores: In this group all the patients perform a 1,5 Tesla RMI. With these data, three methods will be used to calculate the ADC score : Siemens, PACS Carestream, Osirix. The ADC scores obtained with these three post-processing softwares will be compared.
  Interventions: Other: Calculate the ADC scores

INTERVENTIONS:
Other: Calculate the ADC scores — The MRI will be performed on the two groups of patients in the usual care. The intervention will be based on the ADC scores calculation. The scores will be obtained with three types of post-processing softwares : Siemens, PACS Carestream, Osirix.

SUMMARY:
Lumbar spine bone marrow is well explored in Magnetic Resonance Imaging (MRI) but some bone marrow diseases are hard to analyze with this method. Furthermore, there is heterogeneity in normal bone marrow, called apparent diffusion coefficient (ADC). Histological and technical factors appear to be the cause, but the possible influence of the employed post-processing software has never yet been evaluated. The purpose of this study is to determine if there is variability in lumbar bone ADC related to the post-processing software.

DETAILED DESCRIPTION:
Lumbar spine bone marrow is well explored in MRI. Some bone marrow diseases are hard to analyze in conventional MRI, and diffusion-weighted imaging (DWI) could be an additional diagnostic feature. However, according to the literature, there is heterogeneity in normal bone marrow of the quantitative parameter that it provides, called apparent diffusion coefficient (ADC). Histological and technical factors appear to be the cause, but the possible influence of the employed post-processing software has never yet been evaluated. The purpose of this study is to determine if there is variability in lumbar bone ADC related to the post-processing software.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing lumbar spine MRI at University Hospital of Saint-Etienne

Exclusion Criteria:

* <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population studied is composed of 100 patients that will performed an MRI in the CHU de Saint-Etienne. They have lumbar pain, and the MRI is indicated off-study.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2015-11-16 (Actual); Study Completion 2015-11-16 (Actual)

PRIMARY OUTCOMES:
ADC Score according to the post-processing software used | 1 day
  The ADC Score will be calculated for each patient, with three different post-processing softwares : Siemens, PACS (picture archiving and communication system) Carestream, Osirix. The scores will be compared, because the aim of this study is to demonstrate the variability of this score, according to the post-processing software used.
  Apparent diffusion coefficient (ADC) is a measure of the magnitude of diffusion (of water molecules) within tissue, and is commonly clinically calculated using Magnetic resonance imaging (MRI) with diffusion weighted imaging (DWI). An ADC of a tissue is expressed in units of mm2/s. There is no unanimity regarding the boundaries of the range of normal diffusion, but ADC values less than 1.0 to 1.1 x 10-3 mm2/s (or 1000-1100 x 10-6 mm2/s) are generally acknowledged in adults as indicating restriction.

SECONDARY OUTCOMES:
ADC Score according to the intensity of MRI | 1 day
  The ADC Score will also be compared to the intensity of the Magnetic resonance imaging (MRI) performed for each patient. Half have received a MRI of 1,5 Tesla and the other hand a 3 Tesla MRI. The variability between these two groups will be compared in the secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Claire BOUTET, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint Etienne, Saint-Etienne, Saint Priest En Jarez, France

IPD SHARING:
Plan to Share IPD: No